CLINICAL TRIAL: NCT00912626
Title: Family Functioning and Child Behavior When a Sibling is Critically Ill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-2-6426
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2014-04

CONDITIONS: Child Behavior
Keywords: siblings; family; child behavior; critical illness; social support
MeSH Terms: conditions — Child Behavior; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FU-1 feedback (Experimental)
  Interventions: Behavioral: One week follow up assessment results
- control group (No Intervention)

INTERVENTIONS:
Behavioral: One week follow up assessment results — FU-1 feedback group will receive child behavior assessment results and interpretation,and a brief intervention to encourage support options.
  Arms: FU-1 feedback

SUMMARY:
The goal of this study is to determine if there is a correlation between an efficacious family environment and sibling behavior in families with children who are critically ill.

DETAILED DESCRIPTION:
Families of critically ill children can face many emotional challenges during the course of a child's illness. While some research has looked at the impact on parents, there has been little focused on siblings. We want to better understand how social support may have a protective effect on siblings' quality of life. The goal of this study is to determine if there is a correlation between an efficacious family environment and sibling behavior in families with children who are critically ill. Our hypothesis is that a cohesive, emotionally rich and open family environment provides social support so that siblings can explore and express the difficult emotions that accompany illness, and is therefore a protective factor for a sibling's behavior.

ELIGIBILITY:
Inclusion Criteria:

* adult (age 18 and older) who has decision making authority for CHOP patient who has been referred to the Pediatric Advanced Care Team (PACT) for palliative care services, and with a child(ren) age 6-11 years who is a sibling of the patient
* any race/ethnicity

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To compare behavioral assessment scores of siblings of children who are critically ill to scores of the general population | baseline and 6 months

SECONDARY OUTCOMES:
To assess if parents who receive results of sibling behavior scores and a brief intervention, compared to parents who do not receive this information or intervention, have a different perception of the sibling's strengths and difficulties. | baseline and 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Chris Feudtner, MD, PhD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States